

Protocol Number: 20110110 Date: 22 FEBRUARY 2018

## STATISTICAL ANALYSIS PLAN

| Protocol Title: | A Multicenter, Controlled, Open-label Extension (OLE) Study to Assess the Long-term Safety and Efficacy of AMG 145 | |
|---|---|---|
| Short Protocol Title: | An Open-label Extension (OLE) Study to Assess<br>the Long-term Safety and Efficacy of AMG 145 | |
| Protocol Number: | 20110110 | |
| Authors: | PPD | |
| Sponsor: | Amgen Inc. One Amgen Center Drive, Thousand Oaks, CA, 91320, USA | |
| SAP Date: | <u>Document Version</u> | <u>Date</u> |
| | Original (v[1.0]) | 23 Febuary 2012 |
| | Amendment (v [2.0]) | 22 FEB 2018 |



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

## **Table of Contents**

| Tabl | e of Abbrevia | ations | 4 |
|---|---|---|---|
| 1. | Introduction | າ | 6 |
| 2. | <ul><li>2.1 Prin</li><li>2.2 Sec</li></ul> | naryondaryloratory | 6<br>6 |
| 3. | 3.1 Stud | viewdy Designnple Size | 6 |
| 4. | <ul><li>4.1 Prin</li><li>4.2 Sec</li><li>4.3 Exp</li><li>4.4 Safe</li><li>4.5 Pha</li></ul> | points and Baseline Covariates nary Endpoint condary Endpoints condary Endpoints ety Endpoints armacokinetics Endpoints nned Covariates | 7<br>8<br>8 |
| 5. | Hypothesis | | 9 |
| 6. | 6.1 Stud<br>6.2 Der | dy Time Points<br>nographics and Baseline Related Definitionser Study Related Definitions | 10<br>11 |
| 7. | | ubsetsnary Analysis Set | |
| 8. | Interim Ana | alysis and Early Stopping Guidelines | 14 |
| 9. | 9.1 Ger<br>9.2 Data<br>9.3 Har<br>9.3.<br>9.3.<br>9.3.<br>9.4 Deta<br>9.5 Out<br>9.6 Dist | 2 Missing Lipid Panel Endpoint | 14<br>14<br>15<br>15<br>15<br>15<br>16<br>16 |
| 10. | Statistical N | Methods of Analysis | 16 |



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

| | 10.1 | General | l Principles | 16 |
|---|---|---|---|---|
| | 10.2 | Subject | Accountability | 17 |
| | 10.3 | Importa | nt Protocol Deviations | 17 |
| | 10.4 | Demogr | raphic and Baseline Characteristics | 18 |
| | 10.5 | Analyse | es of Primary Endpoint | 19 |
| | | 10.5.1 | General Principles | 19 |
| | 10.6 | Analyse | es of Secondary and Exploratory Endpoints | 20 |
| | | 10.6.1 | Analyses of Secondary Endpoints | 20 |
| | | 10.6.2 | Analyses of Exploratory Endpoints | 20 |
| | | 10.6.3 | Pharmacokinetic or | |
| | | | Pharmacokinetic/Pharmacodynamic Endpoint | 00 |
| | 40.7 | 0-4-4-7 | Analyses | |
| | 10.7 | _ | Analyses | |
| | | 10.7.1<br>10.7.2 | Laboratory Test Results | |
| | | 10.7.2 | Vital SignsAnti-AMG 145 Antibodies | |
| | | 10.7.3 | Exposure to Investigational Product | |
| | | 10.7.4 | Exposure to Other Protocol Specified Treatment | |
| | | 10.7.5 | Exposure to Concomitant Medication | |
| | | 10.7.0 | Steroid Substudy | |
| | | | • | |
| 11. | Chang | ges From | Protocol-specified Analyses | 22 |
| 12. | Literat | ure Citati | ions / References | 23 |
| 13. | Data r | not Cover | ed by This Plan | 24 |
| 14. | Apper | ndices | | 25 |
| | | | List of Tables | |
| T - 1- 1 | . 4 - 1 | | | 4.5 |
| rabi | e 1. Im | putation | Rules for Incomplete Dates | 15 |
| | | | List of Appendices | |
| App | endix A | . Analytic | cal Study Week Assignments | 26 |
| App | endix B | . Commo | on Terminology Criteria for Adverse Events | 29 |
| App | endix C | . Lipid M | odifying Background Therapy | 30 |



Protocol Number: 20110110
Date: 22 FEBRUARY 2018 

## **Table of Abbreviations**

| Abbreviation or Term Definition/Explanation AE Adverse event AHA America Heart Association ApoA1 Apolipoprotein A-1 ApoB Apolipoprotein B AUCt Area under the curve over the dosing interval CEC Clinical Events Committee CHD Coronary Heart Disease Cmax Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
|---|
| AHA America Heart Association ApoA1 Apolipoprotein A-1 ApoB Apolipoprotein B AUCt Area under the curve over the dosing interval CEC Clinical Events Committee CHD Coronary Heart Disease C <sub>max</sub> Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| ApoB Apolipoprotein A-1 ApoB Apolipoprotein B AUCt Area under the curve over the dosing interval CEC Clinical Events Committee CHD Coronary Heart Disease Cmax Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| ApoB Apolipoprotein B AUCt Area under the curve over the dosing interval CEC Clinical Events Committee CHD Coronary Heart Disease Cmax Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| AUCt Area under the curve over the dosing interval CEC Clinical Events Committee CHD Coronary Heart Disease Cmax Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| CEC Clinical Events Committee CHD Coronary Heart Disease C <sub>max</sub> Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| CHD Coronary Heart Disease C <sub>max</sub> Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| C <sub>max</sub> Maximum observed concentration CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| CSR Clinical study report CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| CTCAE NCI Common Terminology Treatment Collaboration ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| ECG Electrocardiogram EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| EOI Events of Interest EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| EOS End of study FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| FAS Full analysis set HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| HDL/LDL RATIO High density lipoprotein/low density lipoprotein ratio |
| HDL-C High density lipoprotein cholesterol |
| HR Heart Rate |
| hsCRP High sensitivity C-reactive protein |
| IBG Independent biostatistical group |
| IC Informed Consent |
| IP Investigational product (AMG 145) |
| IPD Important protocol deviation |
| IVRS Interactive voice response system |
| LDL-C Low density lipoprotein cholesterol |
| Lp(a) Lipoprotein(a) |
| MedDRA Medical dictionary for regulatory activities |
| NCA Noncompartmental analysis |
| NCEP ATP III National Cholesterol Education Panel Adult Treatment Panel III (see References) |
| NYHA New York Heart Association |
| PCSK9 Proprotein convertase subtilisin/kexin type 9 |
| PK Pharmacokinetic |
| PKDM Pharmacokinetics and drug metabolism |
| Q4W Every 4 weeks |
| SC Subcutaneous |



Protocol Number: 20110110 Date: 22 FEBRUARY 2018


| Abbreviation or Term | Definition/Explanation |
|----------------------|------------------------------------------|
| SOC | Standard of care |
| SD | Standard deviation |
| T <sub>max</sub> | Time to maximum observed concentration |
| UC | Ultracentrifugation |
| VLDL-C | Very low density lipoprotein cholesterol |

Protocol Number: 20110110
Date: 22 FEBRUARY 2018 

#### 1. Introduction

The purpose of this statistical analysis plan (SAP) is to provide details of the statistical analyses that have been outlined within the protocol amendment 7 for AMG 145 Study 20110110 – OSLER dated 12 November 2015. The scope of this plan includes the final analysis that are planned and will be executed by the Biostatistics department or designee unless otherwise specified, eg, standard PK tables will be provided by clinical pharmacology modeling and simulation (CPMS).

## 2. Objectives

### 2.1 Primary

To characterize the safety and tolerability of long-term administration of AMG 145

## 2.2 Secondary

Secondary objectives are:

 To characterize the efficacy of long-term administration of AMG 145 as assessed by low density lipoprotein cholesterol (LDL-C) and non-high-density lipoprotein cholesterol (non-HDL-C), apolipoprotein B (ApoB), total cholesterol/HDL-C ratio, and ApoB/Apolipoprotein A-1 (ApoA1) ratio in subjects with hypercholesterolemia

## 2.3 Exploratory

Exploratory objectives are:

- To assess the percent change in fasting plasma lipids (non-HDL-C, apolipoprotein B, total-cholesterol/HDL-C ratio, total cholesterol), and ApoB/ApoA1 ratio, triglycerides, Lp(a), and high sensitivity C-reactive protein (hsCRP)
- To investigate potential biomarker development by biochemical analysis of blood samples
- To characterize pharmacokinetics of AMG 145 and proprotein convertase subtilisin/kexin type 9 (PCSK9) levels
- To estimate cardiovascular event rates in subjects treated with AMG 145 in aggregated exploratory analyses across the AMG 145 program

#### 3. Study Overview

## 3.1 Study Design

This is a multicenter, controlled, open-label extension study to assess the long-term safety and efficacy of AMG 145. Subjects that complete a qualifying protocol will be randomized 2:1 to two treatment groups: Monthly AMG 145 (420mg QM) + standard of care (SOC) or SOC alone for the first year of the study. During the first 12 weeks of the study (blinded post-randomization stabilization period), LDL-C will remain blinded and subjects will remain on the background lipid lowering therapy from the parent study. After 12 weeks, LDL-C will be unblinded and subjects may receive additional



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

lipid-lowering therapy based on local standards of care. Subjects in the SOC only arm will not receive AMG 145 or a placebo injection for the first year of the study.

Randomization should occur at the end of the parent study's end of study (EOS) visit or within 3 days after the parent study's EOS visit and will be stratified by the treatment arm the subject was randomized to in the parent study. Investigators, site staff, subjects, and the study team will be blinded to on-study lipid levels until week 12 (1st quarterly) visit of this study. At the end of the first year (week 52), starting at week 56 (week4/year 2) all subjects will receive open-label AMG 145 for up to 4 years (or until the investigator's recommendation of discontinuation, Amgen's recommendation of discontinuation, the subjects' decision to discontinue for any reason, or until an administrative decision is made to close the study).

## 3.2 Sample Size

The number of subjects entering this study will depend on the number of subjects completing their respective AMG 145 parent studies and willingness to enroll. Approximately 2000 (1970) subjects will be randomized in the qualifying parent studies. Assuming 80% of these subjects enroll in this extension study, the sample size will be approximately 1600 (1576).

The exact 95% confidence intervals for a 5% incidence rate under various enrollment assumptions using the binomial distribution for particular adverse events are provided in the table below. The estimates are derived using SAS version 9.2.

| | Total Number of | Estimated Adverse E | Event Incidence Rate |
|---|---|---|---|
| Percent of Subjects<br>Enrolling | Subjects Reporting Adverse Event | Incidence Rate | 95% Confidence<br>Interval |
| 60 | 59/1182 | 5% | (4%, 6%) |
| 70 | 69/1379 | 5% | (4%, 6%) |
| 80 | 79/1576 | 5% | (4%, 6%) |
| 90 | 89/1773 | 5% | (4%, 6%) |

#### 4. Study Endpoints and Baseline Covariates

## 4.1 Primary Endpoint

Subject incidence of adverse events

## 4.2 Secondary Endpoints

- LDL-C at week 24 and week 52
- non-HDL-C at week 24 and week 52



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

ApoB at week 24 and week 52

- Total cholesterol/HDL-C ratio at week 24 and week 52
- ApoB/ApoA1 ratio at week 24 and week 52

## 4.3 Exploratory Endpoints

- Subject incidence of adjudicated events
  - Death (all cause, cardiovascular)
  - Cardiac ischemic events (myocardial infarction, hospitalization for unstable angina, coronary revascularization)
  - Hospitalization for heart failure
  - Cerebrovascular events (transient ischemic attack, stroke)
- Subject incidence of non-coronary revascularization
- Change and percent change from baseline at each scheduled visit in each of the following lipid parameters:
  - Total cholesterol
  - non-HDL-C
  - LDL-C
  - ApoB
  - total cholesterol/HDL-C ratio
  - ApoB/ApoA1 ratio
  - Triglycerides
  - HDL-C
  - VLDL-C
  - ApoA1
  - Lp(a)
  - hsCRP
- PCSK9 at each scheduled visit

#### 4.4 Safety Endpoints

- Changes from baseline in safety laboratory values (including clinical chemistry and hematology) and vital signs at each scheduled visit
- Subject incidence of anti-AMG 145 antibodies

## 4.5 Pharmacokinetics Endpoints

Serum concentration of AMG 145 at selected time points




Protocol Number: 20110110 Date: 22 FEBRUARY 2018

#### 4.6 Planned Covariates

Covariates include, but not limited to:

### Stratification Factor

- randomized to AMG 145 Q2W in parent study
- randomized to AMG 145 Q4W in parent study
- not randomized to AMG 145 in parent study

## Baseline Covariates from Parent Study

- Demographics
  - age (< 65, ≥ 65)
  - gender
  - race (black, white, and other)
  - region (North America, other)
  - Body Mass Index (BMI) (< 25, 25 < 30, ≥ 30)</li>
  - Weight (< baseline median, ≥ baseline median)</li>
- Medical history
  - diabetes mellitus (yes, no)
  - hypertension (yes, no)
  - current smoker (yes, no)
  - metabolic syndrome per modified AHA/NHLBI criterion (yes, no)
  - baseline CHD risk factors ≥ 2 (yes, no)
  - family history of premature coronary heart disease (yes, no)
- Concomitant medication and laboratory measurement
  - Lipid modifying background therapy (intensive statin usage, non-intensive statin usage, non-statin usage, none [as defined in Appendix D])
  - LDL-C (< baseline median, ≥ baseline median)</li>
  - Triglycerides (< baseline median, ≥ baseline median; < 150 mg/dL,</li>
     ≥ 150 mg/dL, < 200 mg/dL,</li>
  - PCSK9 level (< baseline median, ≥ baseline median)</li>

## 5. Hypothesis

There is no formal hypothesis testing. Subject incidences of adverse events will be estimated.




Protocol Number: 20110110
Date: 22 FEBRUARY 2018


#### 6. Definitions

#### 6.1 Study Time Points

## **Baseline**

Baseline is defined as the parent study baseline.

## First Dose Date

For subjects randomized to AMG 145+SOC, the first dose date is the first date at which the subject was administered IP. For subjects randomized to SOC, the first dose date is the first date at which the subject was administered IP at or after the Week 56 visit.

#### End of Investigational Product (EOIP) Date

If a subject has completed or discontinued IP, the EOIP date is date recorded on the final IP dose date eCRF.

#### End of Study (EOS) Date

For each subject, the end of study date is the date recorded on the End of Study eCRF.

#### **Enrollment Date**

The enrollment date for a subject is either the subject's EOS date for the parent study or the randomization date for Study 20110110, whichever is later.

#### Randomization Date

The randomization date for each subject is the date the investigator (or designee) confirms in the IVRS that the subject has met all eligibility criteria and is randomized.

#### Study Day 1

For subjects randomized to AMG 145 plus SOC arm and received at least one dose of AMG 145, Study Day 1 is defined as the first day that AMG 145 is administered during this study.

For subjects randomized to SOC only arm, or randomized to AMG 145 plus SOC arm but never received AMG 145, Study Day 1 is defined as the randomization date or parent EOS date, whichever is later.

#### Study Day

For each subject, and for a given study visit date, study day is defined as the number of days since Study Day 1:

Study day = (study visit date - Study Day 1 date) + 1

If the date of interest is prior to the Study Day 1:

Study day = (study visit date – Study Day 1 date)



Protocol Number: 20110110
Date: 22 FEBRUARY 2018


#### SOC-Controlled period

The start of the SOC-Controlled period is the Study Day 1.

For end of the SOC-Controlled period:

- If a subject is administered a dose of IP at the Week 56, the day prior to the week 56
   IP date is the end of the SOC-Controlled period.
- If a subject is not administered a dose of IP at Week 56, the SOC-Controlled period will end at the earliest of Study Day 399, and the EOS date.

## All-IP period

Subjects with EOS dates ≤ end of SOC-Controlled period dates will have missing start and end of All-IP period dates.

#### Otherwise:

- All-IP period start date = end of SOC-Controlled period date+1.
- All-IP period end date = EOS date.

#### 6.2 Demographics and Baseline Related Definitions

## Change (absolute change) from Baseline

The arithmetic difference between a post-randomization value and baseline for a given time point: Change from baseline = (post-randomization value – baseline value)

#### Percent Change from Baseline

The percent change from baseline for a given variable at a given time point is defined as: 100 x change from baseline / baseline value

## 6.3 Other Study Related Definitions

#### Analytical Study Week Assignments

Analytical windows will be used to assign parameters to study weeks. The algorithm is provided in Appendix A.

#### IP Exposure Period in Months

IP Exposure Period in months= [(min(EOIP date + 28 days, EOS date) – First dose date) + 1] / 365.25 \* 12. For subjects randomized to SOC treatment during the SOC-Controlled period, the first dose date is equivalent to the first dose date during the All-IP period.



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

#### Study Exposure Period in Months

For each randomized subject, Study Exposure Period in months = [EOS date – enrollment date) + 1] / 365.25 \* 12

## IP Exposure in Months During the SOC-Controlled period

For subjects randomized to AMG 145+SOC arm and received at least one dose of AMG 145 in the SOC-Controlled period, IP Exposure during the SOC-Controlled period = [(min(EOIP date + 28 days, end of SOC-Controlled period) – Study Day 1) + 1] / 365.25 \* 12. Any IP exposure < 0 will be considered as N/A.

For subjects randomized to SOC or randomized to AMG 145 + SOC and not dosed in the SOC-Controlled period, IP Exposure during the SOC-Controlled period = N/A.

### IP Exposure in Months During the All-IP period

For each randomized subject in the Interim All-IP period Analysis Set, IP Exposure during the All-IP period

= [(min(EOIP + 28 days, end of All-IP period) – start date of All-IP period) + 1] / 365.25 \* 12. If the above calculation is < 0, then set to 0.

#### Study Exposure in Months During the SOC-Controlled period

For each randomized subject, Study Exposure Period for the SOC-Controlled period = [(end of SOC-Controlled period date – start of the SOC-Controlled period + 1] / 365.25 \* 12.

#### Study Exposure in Months During the All-IP period

For each randomized subject that received a dose of IP during the All-IP period,

Study Exposure Period for the All-IP period = [(end of All-IP period – start of the All-IP period + 1] / 365.25 \* 12.

## Adverse Events Included in the Summary Tables

An adverse event is included in SOC-Controlled period summaries if it occurs during the SOC-Controlled period and the subject is in the Full Analysis Set.

An adverse event is included in All-IP period summaries if it occurs during the All-IP period and the subject is in the All-IP period Analysis Set.




Protocol Number: 20110110 Date: 22 FEBRUARY 2018

## Baseline Metabolic Syndrome

For each subject without type 2 diabetes mellitus, metabolic syndrome is identified by the presence of 3 or more of the components listed below (modified AHA/NHLBI criteria). Subjects with type 2 diabetes cannot be categorized as having metabolic syndrome.

| Risk Factor | Defining Level |
|---|---|
| Elevated waist circumference: | |
| Non-Asian: | |
| Men | ≥ 102 cm |
| Women | ≥ 88 cm |
| Asian: | |
| Men | ≥ 90 cm |
| Women | ≥ 80 cm |
| Triglycerides | ≥ 150 mg/dL |
| HDL cholesterol | |
| Men | < 40 mg/dL |
| Women | < 50 mg/dL |
| Blood pressure | SBP ≥ 130 mmHg or DBP ≥ 85 mmHg |
| | OR Hypertension checked 'yes' on CV<br>Medical History eCRF |
| Fasting glucose | ≥ 100 mg/dL |

## **4-Level Treatment Group**

All tables in the full analysis set in the final analysis will be summarized by randomization group (AMG 145+SOC vs. SOC alone). Since subjects received either AMG 145 or control treatment in parent study, the tables will be further categorized as the following 4 levels (parent study treatment group/current study treatment group):

"AMG 145/AMG 145 + SOC"; "AMG 145/SOC Only"; "Control/AMG 145 + SOC", and "Control/SOC Only".

#### 7. Analysis Subsets

## 7.1 Primary Analysis Set

#### Full Analysis Set

The full analysis set (FAS) will include all subjects randomized in this study. All analyses of the randomized controlled period of the study will be performed using the FAS. Analyses of the period after the randomized controlled period may be limited to those receiving investigational product.




Protocol Number: 20110110
Date: 22 FEBRUARY 2018

#### The All-IP Period Analysis Set

The All-IP analysis set (AAS) will include all subjects that were randomized in this study and dosed with IP and on-study in the All-IP period. Data will be summarized analyzed from the start of the All-IP period to EOS.

#### Steroid Analysis Set

The steroid analysis set (SAS) includes all subjects who participate in the steroid substudy.

## 8. Interim Analysis and Early Stopping Guidelines

An administrative interim analysis, which included pharmacokinetic / pharmacodynamics (PKPD) modeling and was based on accumulated efficacy and safety data from this and other concurrently conducted studies with AMG 145, was performed by an internal unblinded group to guide future clinical development plans. Members in the designated internal unblinded group did not have direct roles or responsibilities in conducting any study included in this administrative interim analysis. There was an additional 1-year interim analysis to summarize the data collected in the randomized study period (up to week 52) after all subjects had completed the week 52 visits. There were no plans to modify or discontinue this study based on the results of the interim analysis. Also, additional analysis may be performed periodically throughout the study after parent studies are closed and individual subjects are unblinded to their lipid values.

## 9. Data Screening and Acceptance

## 9.1 General Principles

The objective of the data screening is to assess the quantity, quality and statistical characteristics of the data relative to the requirements of the planned analyses.

## 9.2 Data Handling and Electronic Transfer of Data

Amgen's Clinical Data Management department will provide all data to be used in the planned analyses. This study will use the RAVE database.

All data collected in the eCRF will be extracted from RAVE. Protocol deviations will be transferred from eClinical. Details on data transfer will be provided in the Data Transfer Plan.




Protocol Number: 20110110 Date: 22 FEBRUARY 2018

#### 

## 9.3 Handling of Missing and Incomplete Data

#### 9.3.1 Patterns of Missing Data

Subjects may be missing specific data points for various reasons. In general, data may be missing due to a subject's early withdrawal from study, a missed visit, or non-evaluability of a data point or an endpoint at a particular point in time. In the Data Quality Review (DQR) process, queries will be made to the sites to distinguish true missing values from other unknown values (eg, due to measurement or sample processing error). All attempts will be made to capture missing or partial data for this trial prior to the database lock.

The frequency and pattern of missing data for selected endpoints will be assessed through descriptive summaries of the measurements over time.

## 9.3.2 Missing Lipid Panel Endpoint

There will be no imputation for missing lipid panel endpoint.

## 9.3.3 Handling of Incomplete Dates

Adverse event and concomitant medication ([eg, lipid regulatory medication] collected start date data) with completely or partially missing start dates will be queried. After the issue is queried, the date is still incomplete with year only or year and month only, the start date will be imputed as described in Table 1 below.

| | Missing | Imputation | Exception |
|---|---|---|---|
| Start date<br>(AE and | Day | 1st | Default to Study Day 1 if an event starts the same year and month as Study Day 1 |
| concomitant medication) | Day and<br>Month | 1st Jan | Default to Study Day 1 if an event started the same year as Day 1 |

Table 1. Imputation Rules for Incomplete Dates

## 9.4 Detection of Bias

A factor that may bias the results of the study is major protocol deviations likely to impact the analysis and interpretation of the endpoints. Important protocol deviations likely to impact the analysis and interpretation of the endpoints will be tabulated in the Clinical Study Report (CSR).

If any sensitivity analyses are required to evaluate potential biases in the study's conclusions, the sources of the potential biases and results of the sensitivity analyses will be documented in the CSR.



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

#### 9.5 Outliers

Various methods, including univariate summaries, histograms, scatter plots, box plots, and line graphs, may be used to identify outliers in key variables. Extreme data points will be identified during the review of the data prior to database lock. Such data points will be reviewed with clinical data management to ensure accuracy. All analyses will include outliers in the data. Sensitivity analyses may be undertaken if extreme outliers for a variable are observed.

#### 9.6 Distributional Characteristics

There are no distributional requirements for the planned analyses. Therefore no assessment will be made.

## 9.7 Validation of Statistical Analyses

Programs will be developed and maintained, and output will be verified in accordance with current risk-based quality control procedures.

Tables, figures and listings will be produced with validated standard macro programs where standard macros can produce the specified outputs.

The production environment for statistical analyses consists of Amgen-supported versions of statistical analysis software, for example the SAS System and S-plus.

## 10. Statistical Methods of Analysis

#### 10.1 General Principles

Statistical analyses in this open label extension study will be descriptive in nature. No statistical inference is planned.

Subject disposition, demographics and baseline characteristics will be summarized.

Summary statistics for continuous variables will include the number of subjects, mean, median, standard deviation or standard error, 25<sup>th</sup> percentile (Q1), 75<sup>th</sup> percentile (Q3), minimum, and maximum. For categorical variables, the frequency and percentage will be given.

Final analyses will be based on data collected from this study and baseline/some EOS data from the parent studies. Descriptions of any integrated analyses with the parent studies are out of scope for this SAP.

The final analysis will be conducted when all subjects have either completed all the scheduled study visits or have early terminated from the study. At that time, the database will be cleaned, processed and a snapshot will be taken. All endpoints will be




Protocol Number: 20110110 Date: 22 FEBRUARY 2018


analyzed based on this snapshot. For all endpoints, results will be summarized by the treatment group to which subjects are randomized to in this study, unless otherwise specified. Subjects will be further categorized according to whether they were randomized to AMG 145 or not in their parent study. For the SoC-Controlled period, this combined treatment group will have 4 levels (parent study treatment group/year 1 treatment group): "AMG 145/AMG 145 + SOC"; "AMG 145/ SOC only"; "Not AMG 145/AMG 145 + SOC", and "Not AMG 145/SOC only". For the All-IP period, subjects will be further categorized according to year 1 treatment group: "SoC in SoC-Controlled Period/AMG 145 + SOC"; "AMG 145 + SOC in SoC-Controlled Period/AMG 145 + SOC".

Unless specified otherwise, the baseline value is defined as the subject's baseline value from the parent study.

All analyses will be carried out separately for the FAS and the AAS analysis sets, unless specified otherwise. There will be no imputation for missing data. Deaths and major cardiovascular events from this study will be adjudicated by an independent Clinical Events Committee (CEC) to facilitate aggregated analyses across the program. These events adjudicated by the CEC include:

- death by any cause
- cardiovascular death
- myocardial infarction
- hospitalization for unstable angina
- coronary revascularization
- stroke
- hospitalization for heart failure
- transient ischemic attack (TIA)
- non-coronary revascularizations

#### 10.2 Subject Accountability

The number and percent of subjects who were randomized, received IP, completed IP, discontinued investigational product and reasons for discontinuing, completed study, and discontinued study and reasons for discontinuing will be summarized by treatment group and for the SOC-controlled and All-IP periods separately as well as overall.

## 10.3 Important Protocol Deviations

Important Protocol Deviations (IPDs) categories are defined by the study team before the first subject visit and updated during the IPD reviews throughout the study prior to



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

database lock. If a snapshot is being taken during the study rather than a database lock at the end of the study, categories should be updated during the IPD reviews throughout the study prior to database lock. These definitions of IPD categories, sub-category codes and descriptions will be used during the course of the study. The final IPD list is used to produce the Summary of IPDs table (see Section 12.1) and the List of Subjects with IPDs (see Section 12.2).

### 10.4 Demographic and Baseline Characteristics

All baseline tables will be summarized by randomized treatment and for all subjects in the FAS and AAS. Baseline tables will summarize the following: baseline characteristics, demographics, cardiovascular medical history, and laboratory parameters.

All demographics and baseline variables will be populated from the parent studies.

These tables will summarize the following:

- Parent study
- Stratification factor (randomized to AMG 145 Q2W in parent study; randomized to AMG 145 Q4W in parent study; not randomized to AMG 145 in parent study)
- Demographics
  - age (years)
  - age group (< 65, ≥ 65)</li>
  - gender
  - ethnicity
  - race
  - region (North America, Other)
- Characteristics
  - height (cm)
  - weight (kg)
  - body mass index (kg/m²)
- Targeted medical history
  - coronary artery disease (including angina, myocardial infarction [MI], coronary artery bypass graft [CABG], and percutaneous coronary intervention [PCI])
  - cerebrovascular or peripheral arterial disease (including transient ischemic attack [TIA], stroke, carotid or vertebral artery disease, and peripheral arterial disease)
  - atrial fibrillation/flutter (current or former)
  - congestive heart failure (current NYHA class)
  - left ventricular systolic function




Protocol Number: 20110110 Date: 22 FEBRUARY 2018


- cardiac devices/pacemakers
- metabolic syndrome
- CHD risk factors
- Laboratory parameters
  - LDL-C (UC and calculated)
  - Total cholesterol
  - non-HDL-C
  - ApoB
  - Total cholesterol/HDL-C ratio
  - ApoB/ApoA1 ratio
  - Triglycerides
  - Lp(a)
  - ApoA1
  - VLDL-C
  - HDL-C
  - hsCRP
  - PCSK9
  - Vitamin E
  - Steroids
- Lipid-regulating concomitant medications

## 10.5 Analyses of Primary Endpoint

## 10.5.1 General Principles

The Medical Dictionary for Regulatory Activities (MedDRA) version 20.0 or later will be used to code all adverse events (AE) to a system organ class and a preferred term. All analyses will be performed separately for the FAS and AAS analysis sets.

Subject incidence of adverse events, serious AEs, and AEs leading to withdrawal of investigational product, will be tabulated by system organ class and preferred term in descending order of frequency.

Summaries of adverse events and serious AEs occurring in at least 1% of the subjects by preferred term in any treatment arm will be provided in descending order of frequency.

Subject incidence of adverse events associated with injectable protein therapies Hypersensitivity or allergic reactions and potential hepatitis C infections will be summarized by category and preferred term.



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

Subgroup analyses for stratification factor, age group (< 65,  $\geq$  65), sex, and race (if appropriate) will be presented by system organ class and preferred term in descending order of frequency. All races with less than 5% of the total enrolled subjects will be pooled together for summary purposes.

## 10.6 Analyses of Secondary and Exploratory Endpoints

## 10.6.1 Analyses of Secondary Endpoints

The secondary endpoints of percent change and absolute change from baseline will be summarized for each scheduled visit by randomized treatment group in this study and also the combined treatment group (4 levels). All analyses will be performed separately for each of the FAS and AAS analysis sets.

## 10.6.2 Analyses of Exploratory Endpoints

All analyses will be performed separately for the SOC-Controlled period and the All-IP period.

Subject incidence of adjudicated CV endpoints will be summarized. The percent change and change from baseline in laboratory based exploratory endpoints at each scheduled visit will be summarized. For continuous exploratory endpoints, treatment group summary statistics (number of subjects, mean, median, standard deviation or standard error, first and third quartiles, minimum, and maximum) at all scheduled visits will be calculated.

## 10.6.3 Pharmacokinetic or Pharmacokinetic/Pharmacodynamic Endpoint Analyses

Individual and mean serum AMG 145 and PCSK9 concentration-time profiles will be provided using nominal times. Individual and summary statistics of AMG 145 serum concentrations will be provided.

Compartmental exposure-response analyses will not be specified in this analysis plan but will be addressed in *Population Pharmacokinetic and Pharmacodynamic Analysis of AMG 145 in Subjects with Hyperlipidemia Using Data from Amgen Phase 1 and Phase 2 Studies* as a metadata analysis.

These analyses will be performed by the CPMS group.

## 10.7 Safety Analyses

## 10.7.1 Laboratory Test Results

Descriptive statistics will be provided for actual values and changes from baseline in each applicable laboratory parameter at each protocol-specified scheduled visit.




Protocol Number: 20110110 Date: 22 FEBRUARY 2018

Laboratory analytes are provided in the protocol Table 7-1. Lab shift tables using the most current version of the CTCAE version v4.03 (Appendix C) or later grading will be used for the select analytes of interest, when applicable. Shift tables will be provided for the SOC-Controlled period and the All-IP period. The results will be based on the maximum (ie, worst) shift from parent basline to the end of the SOC-Controlled period

## 10.7.2 Vital Signs

Systolic and diastolic blood pressure and heart rate will be summarized using descriptive statistics at each scheduled visit. Summaries will also include the change from baseline at each scheduled visit

#### 10.7.3 Anti-AMG 145 Antibodies

The incidence and percentages of subjects who develop anti-AMG145 antibodies (binding and neutralizing) at any time will be tabulated.

and from the parent baseline to end of the All-IP period, respectively.

## 10.7.4 Exposure to Investigational Product

Descriptive statistics will be produced to describe the patient-month exposure to investigational product, by treatment group for both the FAS and AAS sets as well as overall.

Exposure definitions are provided in Section 6.3.

#### 10.7.5 Exposure to Other Protocol Specified Treatment

The number and proportion of subjects receiving selected lipid regulating medications captured on the Lipid Regulating Concomitant Medications eCRF will be summarized using descriptive statistics. Summaries will be provided for baseline use and use after Study Day 1. The subject incidence of changes in lipid regulating medications during the treatment period will also be provided.

## 10.7.6 Exposure to Concomitant Medication

The number and proportion of subjects receiving the lipid regulating concomitant medications will be summarized by preferred term as coded by the World Health Organization Drug (WHODRUG) dictionary. Summaries will be provided for baseline use and use after Study Day 1.

#### 10.7.7 Steroid Substudy

For steroid summaries, the change will be relative to the week 0 value. Analytes for the steroid substudy (ACTH, FSH, LH, Cortisol, Testosterone, Estradiol) will be summarized for each treatment group using descriptive statistics at each scheduled visit.




Protocol Number: 20110110
Date: 22 FEBRUARY 2018


## 11. Changes From Protocol-specified Analyses

A repeated measures mixed model for the secondary endpoints won't be done in the final analysis because the primary interest of the open label extension study is to characterize the safety and tolerability of long-term administration of AMG 145.

The following analysis won't be done:

Point estimates of group means and their 95% confidence intervals will be presented. Differences in the group means, along with the 95% confidence intervals, of the secondary endpoints will be estimated at each scheduled visit between:

- the AMG 145 + SOC group and the SOC only group in this study, regardless of the treatment arm the subject was randomized to in their parent study, and
- the AMG 145 + SOC group and SOC only group in this study, by whether the subject was randomized to AMG 145 or not in their parent study.



Protocol Number: 20110110
Date: 22 FEBRUARY 2018


#### 12. Literature Citations / References

National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III). Third Report of the National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults (Adult Treatment Panel III) final report. *Circulation*. 2002;106:3143-3421.

Grundy SM et al. Diagnosis and Management of the Metabolic Syndrome: An American Heart Association/National Heart, Lung, and Blood Institute Scientific Statement. *Circulation*. 2005;112:2735-2752.

Alberti KGMM et al. Harmonizing the Metabolic Syndrome: A Joint Interim Statement of the International Diabetes Federation Task Force on Epidemiology and Prevention; National Heart, Lung, and Blood Institute; American Heart Association; World Heart Federation: International Atherosclerosis Society; and International Association for the Study of Obesity. *Circulation*. 2009;120:1640-1645.



Protocol Number: 20110110
Date: 22 FEBRUARY 2018


## 13. Data not Covered by This Plan

Currently there are no pre-planned analyses for the biochemical cardiovascular biomarker objective.



Protocol Number: 20110110
Date: 22 FEBRUARY 2018


14. Appendices



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

## Appendix A. Analytical Study Week Assignments

Selected endpoints will be summarized by scheduled study visits in descriptive analyses. Since the actual visits may not exactly coincide with their scheduled visit day, the actual visit day is mapped to the study visit generally by non-overlapping consecutive intervals covering the entire time continuum, with scheduled visit time being the center of each interval. The mapping intervals for all distinct schedules are summarized in the following table. Week 0 mapping does not pertain to parent study week mapping. Data from the parent studies will use the original analytical weeks in the individual study SAPs.

#### Handling multiple records assigned to an analytical study week:

If there is more than one record in a study week interval, the analytical record for that specific study week will be defined as the record closest to the scheduled study day of that specific study week (7×study week). If two records are equidistant from the scheduled day, then the earlier record will be chosen. If there are multiple records on the same day, the last record will be used.

| Scheduled<br>Visit Week | Vital Signs for<br>AMG 145+SOC group | Vital Signs for SOC only group | Fasting plasma lipids ApoA1, ApoB PCSK9 Chemistry Coagulation Hematology hSCRP, Lp(a) | Anti-AMG 145 antibodies Weight, Physical Exam, Urinalysis |
|---|---|---|---|---|
| Week 4 | (1, 42] | (1, 56] | (1, 56] | (1, 56] |
| Week 8 | (42, 70] | | | |
| Week 12 | (70, 98] | (56, 126] | (56, 126] | (56, 126] |
| Week 16 | (98, 126] | | | |
| Week 20 | (126, 154] | | | |
| Week 24 | (154, 182] | (126, 210] | (126, 210] | (126, 210] |
| Week 28 | (182, 210] | | | |
| Week 32 | (210, 238] | | | |
| Week 36 | (238, 266] | (210, 294] | (210, 294] | (210, 294] |

Page 1 of 2




Protocol Number: 20110110 Date: 22 FEBRUARY 2018

| Da | ~~ | 27 | ۸f | 30 |
|----|----|----|----|----|
| Pa | ue | 21 | OI | วบ |

| | | _ | | ı | |
|---|---|---|---|---|---|
| Scheduled<br>Visit Week | Vital Signs for<br>AMG 145+SOC group | Vital Signs for SOC only<br>group | Fasting plasma lipids ApoA1, ApoB PCSK9 Chemistry Coagulation Hematology hSCRP, Lp(a) | Anti-AMG 145<br>antibodies | Weight, Physical Exam,<br>Urinalysis |
| Week 40 | (266, 294] | | | | |
| Week 44 | (294, 322] | | | | |
| Week 48 | (322, 350] | (294,350] | (294,350] | (294,350] | |
| Week 52 | (350, | (350, | (350, | (350, | (1, End of |
| | End of SOC-Controlled period ] | End of<br>SOC-Controlled<br>period ] | End of SOC-Controlled period ] | End of<br>SOC-Controlled<br>period ] | SOC-Controlled period] |
| Week 56 | [Beginning of<br>All-IP<br>period, 406] | [Beginning of<br>All-IP<br>period, 406] | | | |
| Week 60 | (406, 434] | (406, 434] | | | |
| Week 64 | (434, 462] | (434, 462] | [Beginning of All-IP<br>period,490] | | |
| Week 68 | (462, 490] | (462, 490] | | | |
| Week 72 | (490, 518] | (490, 518] | | | |
| Week 76 | (518, 546] | (518, 546] | (490, 574] | | |
| Week 80 | (546, 574] | (546, 574] | | | |
| Week 84 | (574, 602] | (574, 602] | | | |
| Week 88 | (602, 630] | (602, 630] | (574,658] | | |
| Week 92 | (630, 658] | (630, 658] | | | |
| Week 96 | (658, 686] | (658, 686] | | | |
| Week 100 | (686, 714] | (686, 714] | (658, 742] | | |
| Week 104 | (714,742] | (714,742] | | [Beginning of<br>All-IP<br>period, 910] | |
| Week n | ([n-2]*7,<br>[n+2]*7] | ([n-2]*7,<br>[n+2]*7] | ([m-6]*7, [m+6]*7] | ([q-26]*7,[q+26]<br>*7] | |
| Week 260 | >1806 | >1806 | >1806 | >1638 | ≥Beginning of<br>All-IP period |

Page 2 of 2

#### Note:

 $\begin{array}{l} n=108,112,116,120,124,128,132,136,140,144,148,152,156,160,164,168,172,176,180,\\ 184,188,192,196,200,204,208,212,216,220,224,228,232,236,240,244,248,252,256.\\ m=112,124,136,148,160,172,184,196,208,220,232,244,256\\ q=156,208,260 \end{array}$ 



Protocol Number: 20110110 Date: 22 FEBRUARY 2018

| Page 28 of 3 | 30 |
|--------------|--------|
| | $\neg$ |

| Scheduled Visit Week | Vitamin E | Steroids |
|---|---|---|
| Week 0 | ≤1 | ≤1 |
| Week 12 | (1,126] | (1,126] |
| Week 24 | (126,266] | (126,266] |
| Week 52 | (266, End of SOC-Controlled period] | (266, End of SOC-Controlled period] |
| Week 76 | [Beginning of All-IP period, 616] | |
| Week 100 | (616,728] | |

Protocol Number: 20110110 Date: 22 FEBRUARY 2018

## **Appendix B. Common Terminology Criteria for Adverse Events**

Refer to the NCI Common Terminology Criteria for AEs (CTCAE) Version 4.0, published: May 28, 2009 (v4.03: June 14, 2010) for AE and lab shift grading and information. The CTCAE is available at the following link:

http://evs.nci.nih.gov/ftp1/CTCAE/About.html




Protocol Number: 20110110 Date: 22 FEBRUARY 2018

# Appendix C. Lipid Modifying Background Therapy Based on ACC/AHA guidelines:

| | HIGH-INTENSITY<br>STATIN THERAPY | MODERATE-INTENSITY<br>STATIN THERAPY | LOW-INTENSITY<br>STATIN<br>THERAPY | Notes (classification of atypical doses) |
|---|---|---|---|---|
| Atorvastatin | 40 mg or greater<br>QD | 10 mg QD up to less<br>than 40 mg QD | Less than 10 mg<br>QD | Atorvastatin 30 mg<br>QD is Moderate<br>intensity. |
| Rosuvastatin | 20 mg or greater<br>QD | 5 – < 20 mg QD | less than<br>5 mg QD | Rosuvastatin < 5 mg QD is low intensity , Rosuvastatin 15 mg QD = moderate |
| Simvastatin | 80 mg or greater<br>QD | 20-80 mg QD | < 20 mg QD | And Simvastatin > 40 and < 80 mg QD is moderate, Simvastatin 80 mg or greater QD = high, Simvastatin < 20 mg QD is low-intensity |
| Pravastatin | | 40 mg or greater QD | less than<br>40 mg QD | Pravastatin < 10 mg<br>QD is low intensity |
| Lovastatin | | 40 mg or greater QD | less than<br>40 mg QD | Lovastatin 80 mg<br>QD = moderate,<br>Lovastatin 10 mg<br>QD = Low-intensity |
| Fluvastatin | | 80 mg QD | less than<br>80 mg QD | Fluvastatin 10 mg<br>QD = Low-intensity |
| Pitavastatin | | ≥ 2 mg QD | < 2 mg QD | |

UNKNOWN-INTENSITY STATIN THERAPY if dose frequency is other or dose unit is other and therefore total daily dose in mg cannot be derived; NO STATIN THERAPY if subject does not use any statin at baseline.

